CLINICAL TRIAL: NCT01226173
Title: Study of Bio-Rad Laboratories Platelia Dengue NS1 Ag Assay in Blood Donors.
Brief Title: Dengue Virus NS1 Antigen (Bio-Rad) Clinical Protocol
Status: Completed | Type: Observational
Sponsor: Bio-Rad Laboratories (Industry)
Collaborators: American National Red Cross (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ARC IRB Protocol # 2009-037; 1RC2HL101632-01 (NIH)
Record Dates: First submitted 2010-10-19; First posted 2010-10-22 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Mass Screening
Keywords: Prospective screening of blood donors.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA plasma samples contained in plasma preparation tubes (PPTs) that have been frozen within 24 hours of collection and following centrifugation (under the same centrifugation conditions as used for PPTs used for nucleic acid testing, NAT) will be the primary samples for prospective testing.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bio-Rad Platelia Dengue NS1 Ag test — The purpose of the study is to screen blood donors for the presence of dengue NS1 antigen at the ARC in Puerto Rico region using the Bio-Rad Platelia Dengue NS1 Ag test.

SUMMARY:
The purpose of the study is to screen blood donors for the presence of NS1 antigen of the dengue virus at the American Red Cross in Puerto Rico region (and Monroe County, Florida) using the Platelia Dengue NS1 Ag enzyme immunoassay.

DETAILED DESCRIPTION:
Dengue is an endemic disease that is increasingly more common in tropical climates and the dengue epidemic in Puerto Rico (May 2009) presents a risk to the blood supply in Puerto Rico. Also, on July 13th 2010 federal officials reported an outbreak of dengue fever in Florida after a survey of Key West residents found that at least 5% had been infected or exposed to the virus. Therefore this IND study is being carried out to identify blood donors carrying the dengue virus using the Platelia Dengue NS1 Ag (Bio-Rad, France). Prospective testing is being performed on blood donors who have read an information sheet regarding the use of donated blood samples in research. Testing will occur at the American Red Cross, Charlotte, NC NTL site.

ELIGIBILITY:
Inclusion Criteria:

The Puerto Rico Region and Monroe County, Florida will maintain a log of all blood donors enrolled by collection date documenting the time of collection, centrifugation and freezing; only centrifuged and frozen PPTs will be sent to the Charlotte NTL for NS1 Ag testing. Samples frozen when received at the Charlotte NTL will be tested. Samples that arrive thawed will be tested if the time unfrozen is 24 hours or less. When necessary, alternate PPTs (surplus samples used for NAT) will be used for dengue NS1 Ag testing; a log will be kept by the Charlotte NTL documenting the sample identification numbers of thawed samples, approximate time unfrozen and the samples that require an alternate PPT for dengue NS1 Ag testing.

Exclusion Criteria:

Samples that are deemed unacceptable for testing include those held for excessive storage times when thawed (in excess of 24 hours unfrozen or otherwise as determined by the Principal Investigator) or that are cracked or otherwise damaged. Samples having inadequate volume for initial and repeat testing in duplicate will not be tested as determined by the Charlotte NTL; a log will be kept of samples unacceptable for testing and the reason that the samples are unsuitable for testing.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The initiation of the dengue NS1 Ag IND study began on March 8th, 2010 with a study population of donations collected by the American Red Cross in Puerto Rico and the study population was expanded to Monroe County blood collections of the Community Blood Centers of Florida, Inc in August 2010. Testing of collections may be further expanded to include other non-ARC sites in Puerto Rico, or to sites in the continental US with documented local dengue virus transmission. Testing may also include retrospective testing of a repository of samples retained from Puerto Rico during the 2009 epidemic season.Testing will be performed from donors who have read information sheets specific to this study (Dengue Research Study Donor Information).
Sampling Method: Non-Probability Sample
Enrollment: 182353 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of blood donors with repeatedly reactive Platelia Dengue NS1 Ag test results. | Two and a half years
  Platelia Dengue NS1 Ag test results on blood donors at the specified locations will be recorded and reported. Any donation with a reactive or Not Tested result will be placed on Hold until it is confirmed that the region has applied the appropriate deferral assertion on the donor.

SECONDARY OUTCOMES:
Number of blood donors with PCR and/or TMA confirmed positive dengue test results. | Two and a half years
  Platelia Dengue NS1 Ag test results on retrieved plasma units of repeatedly reactive blood donor samples will be recorded, also confirmatory testing (PCR and /or TMA test results) for these blood donors samples will be recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stramer, PhD, Principal Investigator — American National Red Cross
Locations (2):
- Community Blood Centers of Florida, Inc., Lauderhill, Florida, United States
- American Red Cross, San Juan, Puerto Rico

REFERENCES:
- [Background] Dussart P, Labeau B, Lagathu G, Louis P, Nunes MR, Rodrigues SG, Storck-Herrmann C, Cesaire R, Morvan J, Flamand M, Baril L. Evaluation of an enzyme immunoassay for detection of dengue virus NS1 antigen in human serum. Clin Vaccine Immunol. 2006 Nov;13(11):1185-9. doi: 10.1128/CVI.00229-06. Epub 2006 Sep 20. PMID 16988003
- [Background] Bessoff K, Phoutrides E, Delorey M, Acosta LN, Hunsperger E. Utility of a commercial nonstructural protein 1 antigen capture kit as a dengue virus diagnostic tool. Clin Vaccine Immunol. 2010 Jun;17(6):949-53. doi: 10.1128/CVI.00041-10. Epub 2010 Apr 21. PMID 20410325
- [Background] Kumarasamy V, Chua SK, Hassan Z, Wahab AH, Chem YK, Mohamad M, Chua KB. Evaluating the sensitivity of a commercial dengue NS1 antigen-capture ELISA for early diagnosis of acute dengue virus infection. Singapore Med J. 2007 Jul;48(7):669-73. PMID 17609831
- [Background] Alcon S, Talarmin A, Debruyne M, Falconar A, Deubel V, Flamand M. Enzyme-linked immunosorbent assay specific to Dengue virus type 1 nonstructural protein NS1 reveals circulation of the antigen in the blood during the acute phase of disease in patients experiencing primary or secondary infections. J Clin Microbiol. 2002 Feb;40(2):376-81. doi: 10.1128/JCM.40.02.376-381.2002. PMID 11825945